CLINICAL TRIAL: NCT00230529
Title: A Phase II, Multicenter, Randomized, Double-blind, Placebo-controlled Trial Evaluating the Efficacy and Safety of Infliximab (REMICADE�) Induction Therapy in Patients With Plaque-type Psoriasis
Brief Title: A Safety and Efficacy Study of Infliximab (Remicade) in Patients With Plaque Type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003124; NCT01128491 (obsolete NCT alias)
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2010-08

CONDITIONS: Psoriasis
Keywords: Plaque-type Psoriasis; infliximab; Remicade; biologics
MeSH Terms: conditions — Psoriasis | interventions — Infliximab

INTERVENTIONS:
Drug: infliximab

SUMMARY:
The purpose of the study is to evaluate the effectiveness and safety of infliximab (Remicade) in patients with plaque-type psoriasis.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the safety and possible usefulness of infliximab therapy for patients with severe plaque psoriasis. In a previous small study of infliximab in 33 patients with psoriasis, about 80% of patients treated with infliximab showed improvement in their psoriasis symptoms after the first 3 infusions, while 20% of patients who received placebo showed improvement. The patients will receive infusions of infliximab either 3 or 5 mg/kg or placebo at weeks 0,2,6. Patients who have significant psoriasis at week 26 will receive an additional infusion.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older at time of enrollment
* may be male or female
* Have had a diagnosis of plaque-type psoriasis at least 6 months prior to screening
* Have plaque-type psoriasis covering at least 10% of total BSA at baseline
* Have previously received PUVA and/or other systemic treatment for psoriasis

Exclusion Criteria:

* Have non-plaque forms of psoriasis
* Have a history of drug-induced psoriasis
* Are pregnant, nursing, or planning pregnancy within 12 months of enrollment
* Have had any previous treatment with infliximab or any therapeutic agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving a = 75% improvement in PASI score from baseline at week 10

SECONDARY OUTCOMES:
The proportion of patients positive for antibodies to infliximab;The proportion of patients with infusion reactions at week 26;The proportion of infliximab-treated patients with infusion reaction at week 26 by antibodies to infliximab status at week 26

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Result] Gottlieb AB, Evans R, Li S, Dooley LT, Guzzo CA, Baker D, Bala M, Marano CW, Menter A. Infliximab induction therapy for patients with severe plaque-type psoriasis: a randomized, double-blind, placebo-controlled trial. J Am Acad Dermatol. 2004 Oct;51(4):534-42. doi: 10.1016/j.jaad.2004.02.021. PMID 15389187
- [Result] Feldman SR, Gordon KB, Bala M, Evans R, Li S, Dooley LT, Guzzo C, Patel K, Menter A, Gottlieb AB. Infliximab treatment results in significant improvement in the quality of life of patients with severe psoriasis: a double-blind placebo-controlled trial. Br J Dermatol. 2005 May;152(5):954-60. doi: 10.1111/j.1365-2133.2005.06510.x. PMID 15888152
- See also: A Phase II, Multicenter, Randomized, Double-blind, Placebo-controlled Trial Evaluating the Efficacy and Safety of Infliximab (REMICADE�) Induction Therapy in Patients with Plaque-type Psoriasis. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=142&filename=CR003124_CSR.pdf